CLINICAL TRIAL: NCT06146894
Title: The Effect of Different Obturation Techniques on Postobturation Pain in Single-Visit Root Canal Treatment: A Prospective Clinical Randomized Study
Brief Title: The Effect of Different Obturation Techniques on Postobturation Pain in Single-Visit Root Canal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hisham Mahmoud Hamdy Abada, Doctor, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HA2427
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Bioceramic sealer; Obturation
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single cone technique (Bioceramic Sealer) (Experimental)
  Interventions: Procedure: Single obturation technique (Bioceramic Sealer)
- lateral condensation technique (Bioceramic Sealer) (Experimental)
  Interventions: Procedure: lateral condensation technique (Bioceramic Sealer)
- Warm Vertical condensation technique (Bioceramic Sealer) (Experimental)
  Interventions: Procedure: Warm Vertical condensation technique (Bioceramic Sealer)
- lateral condensation technique (AH plus Sealer) (Experimental)
  Interventions: Procedure: lateral condensation technique (AH Plus Sealer)
- Warm Vertical condensation technique (AH plus Sealer) (Experimental)
  Interventions: Procedure: Warm Vertical condensation technique (AH plus Sealer)

INTERVENTIONS:
Procedure: Single obturation technique (Bioceramic Sealer) — Root canal will be obturated using single cone technique using Bioceramic Sealer
  Arms: Single cone technique (Bioceramic Sealer)
Procedure: lateral condensation technique (Bioceramic Sealer) — Root canal will be obturated using lateral condensation technique using Bioceramic Sealer
  Arms: lateral condensation technique (Bioceramic Sealer)
Procedure: Warm Vertical condensation technique (Bioceramic Sealer) — Root canal will be obturated using vertical condensation technique using Bioceramic Sealer
  Arms: Warm Vertical condensation technique (Bioceramic Sealer)
Procedure: lateral condensation technique (AH Plus Sealer) — Root canal will be obturated using lateral condensation technique using AH plus Sealer
  Arms: lateral condensation technique (AH plus Sealer)
Procedure: Warm Vertical condensation technique (AH plus Sealer) — Root canal will be obturated using vertical condensation technique using AH plus Sealer
  Arms: Warm Vertical condensation technique (AH plus Sealer)

SUMMARY:
The goal of this prospective clinical randomized study is to evaluate the effect of different obturation techniques on postobturation pain in single-visit root canal treatment in 18-60 years old patient who present no systemic disease (American Society of Anesthesiology class I or II) and require nonsurgical root canal treatment The main question it aims to answer which obturation technique used with bioceramic sealer cause less postobturation pain in single-visit root canal treatment in comparison to AH plus sealer used with lateral condensation or warm vertical compaction.

Participants will receive single visit root canal treatment using bioceramic sealer with different obturation techniques Group 1: Single cone technique Group 2: lateral condensation technique Group 3: Vertical compaction technique to see effect of different obturation technique on postobturation pain in single-visit root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years who presented no systemic disease (American Society of Anesthesiology class I or II) and required nonsurgical root canal treatment.
* Diagnosis of asymptomatic irreversible pulpitis in a molar tooth with 3 independent root canals.

Exclusion Criteria:

* Presence of immature root apexes, root fracture, or periodontal disease
* Use of any analgesic, anti- inflammatory, or antibiotics before the treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
postobturation pain | 30 days
  Presence of post-obturation pain will accessed by visual analog scale (VAS) scale (0-10), where 0 showed no pain, 1-3 mild pain, 4-6 moderate pain, 7-9 severe pain, and 10 worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Abada, PhD, Principal Investigator — Kafrelsheikh University
Locations (1):
- kafrelsheikh University, Kafr ash Shaykh, Kafr El-Shaikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36385378/